CLINICAL TRIAL: NCT06584240
Title: A Phase Ib/II Clinical Study to Evaluate the Safety and Efficacy of Recombinant Botulinum Toxin Type A (JHM03) in Adult Patients With Upper Limb Spasticity
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of JHM03 in Adult Patients With Upper Limb Spasticity
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: JHM BioPharma (Tonghua) Co. , Ltd. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JHM03-CT102
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Upper Limb Spasticity

STUDY DESIGN:
Intervention Model Description: JHM03 and Placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Experimental Group 1 (Experimental): Participants will receive one cycle of JHM03 in the selected overactive upper limb muscles
  Interventions: Drug: Sequence 1
- Experimental Group 2 (Experimental): Participants will receive one cycle of JHM03 in the selected overactive upper limb muscles
  Interventions: Drug: Sequence 2
- Experimental Group 3 (Experimental): Participants will receive one cycle of JHM03 in the selected overactive upper limb muscles
  Interventions: Drug: Sequence 3
- Experimental Group 4 (Experimental): Participants will receive one cycle of JHM03 in the selected overactive upper limb muscles
  Interventions: Drug: Sequence 4
- Placebo Group (Placebo Comparator): Participants will receive one cycle of Placebo in the selected overactive upper limb muscles
  Interventions: Drug: Sequence 5

INTERVENTIONS:
Drug: Sequence 1 — Single treatment, intramuscularly injected. The total injection 100-150U.
  Arms: Experimental Group 1
Drug: Sequence 2 — Single treatment, intramuscularly injected. The total injection 200-250U.
  Arms: Experimental Group 2
Drug: Sequence 3 — Single treatment, intramuscularly injected. The total injection 350-400U.
  Arms: Experimental Group 3
Drug: Sequence 4 — Single treatment, intramuscularly injected. The total injection ≤400U.
  Arms: Experimental Group 4
Drug: Sequence 5 — Single treatment, intramuscularly injected.
  Arms: Placebo Group

SUMMARY:
This is a phase Ib/II clinical study to evaluate the safety and efficacy of recombinant botulinum toxin type A（JHM03）in adult patients with upper limb spasticity. The purpose of this study was to observe efficacy and safety of JHM03 compared with placebo in adult patients with upper limb spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 80 years of age inclusive, at the time of signing the informed consent
* Body weight ≥50Kg
* Participants with stable post-stroke Spasticity (ULS) for at least 3 months
* Participants with Modified Ashworth Scale (MAS) score of at least 2 at elbow flexor or wrist flexor or finger flexor
* Participants with DAS score of at least 2 on the Principal Target of Treatment (PTT) (one of four functional domains: dressing, hygiene, limb position and pain)
* Participants who have been stable for at least 1 month prior to study entry in terms of oral antispasticity

Exclusion Criteria:

* Previous use of any botulinum toxin within 6 months prior to screening, or plan to use any botulinum toxin during the study.
* History of alcohol or drug abuse.
* Known allergy or hypersensitivity to any component of the study products.
* History of epilepsy
* Known or suspected to be HIV positive, serologically positive for syphilis, or active hepatitis B or C
* Any medical condition that may put the participant at increased risk for botulinum toxin type A use

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-05-24 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
The incidence rate of adverse events and severe adverse events | Within 12 weeks
  The incidence rate of adverse events and severe adverse events within 12 weeks after injection;
Change from baseline at week 4 for primary targeted muscle group on the MAS | Within 4 weeks
  Change from baseline at week 4 for primary targeted muscle group on the MAS(Modified Ashworth Scale).

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Beijing Tsinghua Changgung Hospital, Beijing, Beijing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Huazhong University of Science and Technology Union Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical Hospital, Shijiazhuang, Hebei
  - Luoyang Central Hospital, Luoyang, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Huai 'an Second People's Hospital, Huai'an, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning
  - Rizhao People's Hospital, Rizhao, Shandong
  - Yantai Mountain Hospital, Yantai, Shandong
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Yangzhi Affiliated Rehabilitation Hospital of Tongji University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No